CLINICAL TRIAL: NCT03878797
Title: An Observational Study of The Depth of Endotracheal Tube Insertion
Brief Title: The Depth of Endotracheal Tube Insertion
Status: Completed | Type: Observational
Sponsor: Gao Mei (Other)
Responsible Party: Sponsor-Investigator, Gao Mei, Assistant Director, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Other Study IDs: 2019-SR-041
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Endotracheal Intubation
Keywords: Endotracheal tube; Endobronchial intubation; Vocal cords; Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

SUMMARY:
Virtual experiment : comparing the new method with conventional method of determining the depth of endotracheal intubation.

DETAILED DESCRIPTION:
Effective airway management is the primary concern of the anesthesiologist. The conventional method of determining the insertion length of the endotracheal tube, 21 cm for women and 23 cm for men, shows a high incidence of endobronchial intubations in the analyzed population.The aim of this study is form a new and safe practice habit by passing the endotracheal tube with the balloon just 2 cm below the vocal cords during intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for elective surgery under general anesthesia

Exclusion Criteria:

* Patients with anatomical defects of the face, neck, or upper airway
* Patients at risk for pulmonary aspiration of gastric content

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: adult patients who are scheduled for elective surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
the depth of primary insertion of tracheal tube | in a minute after intubation

SECONDARY OUTCOMES:
the distance from the corner of mouth to the carina | in a minute after intubation
the distance from the vocal cords to the carina | in a minute after intubation
the distance from the corner of mouth to the vocal cords | in a minute after intubation

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided